CLINICAL TRIAL: NCT03465228
Title: Effects of Photobiomodulation and Deep Water Running Training in Subjects With Low Back Pain: a Randomized Controlled Trial
Brief Title: Effects of Photobiomodulation and Deep Water Running Training in Subjects With Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Universidade Estadual de Maringá (Other)
Responsible Party: Principal Investigator, Rodrigo Antonio Carvalho Andraus, Doctor, Universidade Norte do Paraná
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 87013
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain; Hydrotherapy; Exertion; Excess
Keywords: Low Back Pain; Photobiomodulation; Deep Water Running; Training; Running
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The first day, will be explanation of the project and signing of the Informed Consent Term. The participants will go to collect blood samples for analysis creatine kinase and cortisol levels. They will be submitted an anthropometric evaluation, psychometric questionnaires and perform functional tests, and perform of a continuous submaximal exertion test. All these procedures will be performed again at the end of the intervention, and the pain intensity scale will be applied in all meetings with participants (beginning and end of each session). After the evaluations, the participants will be randomized into three experimental groups with 15 participants in each: the first group will be the training group that will perform interval training sessions in addition to continuous training sessions. The second group will perform the same training model, and before the training sessions the LED will be applied. And the third group will only receive the LED application.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be not informed if the LED appliance will be on or off, and the outcomes will be numbers for identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Training group (Experimental): This group will do the Deep Water Running, with intervals and continuous training twice a week, and before each session, will be applied the LED equipment. The training will be thirty minutes and will be controlled by heart rate, 70% to 80% maximum heart rate in continuous training, and maximum heart rate in intervals training.
  Interventions: Device: Training group
- Training and LED group (Experimental): This group will receive the photobiomodulation treatment and the same training model of training group.
  Interventions: Device: Training and LED group; Device: Training group
- LED group (Experimental): This group will receive only the photobiomodulation treatment with 30 seconds of light emitting in four points of lumbar region.
  Interventions: Other: LED group

INTERVENTIONS:
Device: Training and LED group — The LED application will be performed before GTL training sessions and will be applied through the spot method with direct contact of the equipment over the irradiated site for 30 seconds. The application will be in four points in the lumbar region, above the gluteal region, with an angle of 90 ° in relation to the cutaneous surface. A wavelength of 660 to 850nm will be used with a frequency of 0 to 1500 Hz and energy irradiated of 0.9 J of each diode totaling 43.2J (48 diodes).
  Arms: Training and LED group
Device: Training group — The training sessions will be monitored based on the subjective perception of exertion of the session (PSESession) (FOSTER, 1998), and heart rate. There will be two types of training: continuous and interval training. The sessions of the training group (GT) and group training + LED (GL) will be preceded by a warm-up of 15 minutes. Participants in the two training groups will undergo weekly training twice weekly on non-consecutive days during four weeks. Continuous training will be 30 minutes at 70% to 80% of maximum heart rate, and interval training will be performed 30 minutes at 100% maximum heart rate of laced racing with fixation of an elastic tube in the floating vest, 30 seconds of intense running and 30 seconds interval. The LED off will be performed before training sessions.
  Arms: Training and LED group; Training group
Other: LED group — This group will be applied through the spot method with direct contact of the equipment over the irradiated site for 30 seconds. The application will be in four points in the lumbar region, above the gluteal region, with an angle of 90 ° in relation to the cutaneous surface. A wavelength of 660 to 850nm will be used with a frequency of 0 to 1500 Hz and energy irradiated of 0.9 J of each diode totaling 43.2J (48 diodes).
  Arms: LED group

SUMMARY:
Physical exercises proves to be an option to revert a vicious cycle and aggravation of the painful that chronic low back pain can provide, which can improve the mobility and stabilization of the spine, muscle strength, motor coordination and general aerobic conditioning. In addition, photobiomodulation using light emitting diodes (LEDs) has attracted attention for acute and chronic pain and wound healing, being used as a resource for prevention and recovery of lesions. Thus, the present study aims to analyze the efficacy of aerobic training systematized with Deep Water Running associated with photobiomodulation in individuals with chronic nonspecific low back pain. Individuals of both sexes, sedentary, who present chronic low back pain, aged between 30 and 55 years (middle-aged individuals) who meet the inclusion and exclusion criteria will be invited to participate. Anthropometric measurements, maximal stress test, functional tests, physiological measures and questionnaires concerning disability and pain, besides psychological ones, will be carried out. After the evaluations, the participants will be randomized into three experimental groups with 15 participants in each: the first group will be the training group that will hold interval training sessions in addition to continuous training sessions (GT). The second group will perform the same training model, and before the training sessions the LED will be applied (GTL). And the third group will only receive the LED application (GL).

DETAILED DESCRIPTION:
This study will be a randomized clinical trial, structured according to the Consort-Statement, with a standardization that includes methodological design, conduction, analysis and interpretation and evaluation of results. The participants will be individuals of both sexes, sedentary, who present chronic low back pain, aged between 30 and 55 years (middle-aged individuals), will be invited to participate. Participants will be informed of all experimental procedures of the study and will sign the Informed Consent Form and to answer the socio-demographic questionnaire. Participation in the study will be voluntary and free of any bonuses or liens; all participants will be free to withdraw their consent at any time without any loss. Prior to the tests, participants will perform prior clinical examinations with the cardiologist to have their cardiac fitness and release checked to carry out the pertinent evaluations of the study. The possible discomfort felt after the tests and training such as tiredness, muscular pain, perspiration will be similar to the senses during the practice of physical exercises. The procedures to be used in this research will follow the regulations required in Resolution 196/96 of the National Health Council on research involving human beings.

Evaluation protocol Body mass index and skin folds of triceps, subscapular, pectoral, abdominal, thigh mean, suprailiac and mean axillary for subsequent determination of fat percentage.

6-minute walk test-adapted The 6-minute walk test consists of a test that evaluates the distance a person can walk on a flat, rigid surface in six minutes and has as main goal the determination of exercise tolerance and oxygen saturation during a submaximal exercise . This test will be adapted to aquatic environment (CAMARGO et al., 2009).

Sit-up test The sit-up test, which consists of quantifying how many supports (hands and / or knees or, still, hands or forearms on knees), the individual uses to sit and lift from the floor. This method of evaluation allows us to analyze items such as flexibility of the lower limb joints, balance, motor coordination and the relation between muscular power and body weight, which can be characterized as minimum functional muscular fitness (ARAUJO, 1999).

Schober's Test To measure the range of motion of the lumbar spine, the Schober test will be performed, which consists of placing a tape measure from the lumbosacral joint, 10 cm above with the individual in a neutral position, and request the trunk flexion, where the increase of the distance between the marks will provide the estimate of the flexion amplitude of the lumbar spine (Schober, 1937).

Determination of cortisol and creatine kinase's blood markers At the beginning and at the end of the training period, blood samples will be collected for the determination of creatine kinase and cortisol levels. They will be stored in Eppendorf and then centrifuged at 3000rpm for 10 min. Serum will be stored at -20⁰C, while plasma will be discarded, and it wil be read with ck and cortisol analysis kit.

Determination of mood, disability, pain intensity Questionnaires will be applied to monitor the state of beliefs and fears, disability and intensity of pain. The Fear avoidance beliefs questionnaire (FABQ) questionnaire, an instrument for assessing the beliefs and fears of individuals with low back pain and how this pain may affect their physical activities, FABQ-Phys subscale, and occupational subscale, subscale FABQ-Work. It consists of 16 self-report items, which are divided into two subscales: the one that addresses the fears and beliefs of individuals in relation to work and in relation to physical activities. Each item is graded on a seven-point scale, ranging from 0 (completely disagree) to 6 (completely agree) (ABREU et al., 2008), and will be applied at the baseline and after the interventions are completed.

The Oswestry Questionnaire presents 10 sections describing pain or limitations resulting from low back pain, The Oswestry Questionnaire presents 10 sections describing pain or limitations resulting from low back pain, will be applied before and after the intervention period. Each section presents six items, where the zero score indicates little or no pain and / or functional limitation, while score 5 is indicative of extreme pain and / or limitation (VIGATTO, ALEXANDRE and FILHO, 2007).

To evaluate pain intensity, the EVA (COSTA, et al., 2008), which consists of a subjective evaluation of 0 (no pain) to 10 (lots of pain), will be applied in all sessions before and at the end of it. And for a more careful assessment of pain, McGill (PIMENTA and TEIXEIRA, 1996), which is an instrument that provides quantitative information on pain and allows an association with sensorial, affective and evaluative qualities of the process which will be applied at the beginning and at the end of the interventions.

TRAINING PROTOCOL The training sessions will be monitored based on the subjective perception of effort of the session (FOSTER, 1998), and heart rate. There will be two types of training: continuous and hight intensity interval. The sessions of the training group and group training + LED will be preceded by a warm-up of 15 minutes. Participants in the two training groups will undergo weekly training twice weekly in non-consecutive days during the four week period. A total of four continuous training sessions and four high intensity interval training sessions will be held. Continuous training will be 30 minutes at 70 - 80% HRmax, and interval training will be performed 30 minutes high intensity of laced running with fixation of an elastic tube in the floating vest, 30 seconds intense run in maximum effort and 30 seconds of interval.

LED Application The LED application will be performed in the GL and immediately after the GTL training sessions, and will be applied through the spot method with direct contact of the equipment over the irradiated site for 30 seconds. The application will be in the lumbar region, above the gluteal region, with an angle of 90 ° in relation to the cutaneous surface. A wavelength of 660 to 850 nm will be used with a frequency of 0 to 1500 Hz and energy irradiated of 0.9 J of each diode totaling 43.2J (48 diodes).

ELIGIBILITY:
Inclusion Criteria:

* sedentary
* nonsmoker
* diabetic
* hipertensive
* asthmatic
* cardiovascular disease
* any restriction to the practice of physical exercise
* severe spinal diseases
* previous surgery on the spine
* nerve root compression
* infection or skin lesion at the site of the LED application
* who has been under physiotherapy for chronic low back pain in the last six months

Exclusion Criteria:

* fear of swimming pool
* minimum frequency of 90%
* Unable to finalize training protocol

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Cortisol levels | six weeks
  nmol/L

SECONDARY OUTCOMES:
Visual Analogue Scale - pain intensity | six weeks
  The Visual Analogue Scale - VAS consists of assisting in the measurement of pain intensity in the patient, where 0 means total absence of pain and 10 the maximum level of pain that the patient can bear.
Aerobic performance | six weeks
  meters
Oswestry Disability Index - disability | six weeks
  The Oswestry Disability Index (ODI) is an index for to quantify disability for low back pain. This questionnaire contains ten topics followed by 6 statements describing different potential scenarios in the patient's life. Each question has a scale of 0-5 where the scores for all questions answered are summed, then multiplied to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
McGill Pain Questionnaire - Subjective pain measurement | six weeks
  McGill Pain Questionnaire is a scale of rating pain that describe the quality and intensity of pain that the pacient are experiencing. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Fear-Avoidance Beliefs | six weeks
  FABQ measures patients' fear of pain and his avoidance of physical activity because of their fear. They are 16 items, with each item scored from 0-6 where higher scores on the FABQ are indicative of greater fear and avoidance beliefs.
Functional test (Physical ability) | six weeks
  Index by Sit-up test: this test consists in quantifying how many supports (hands and / or knees or, still, hands or forearms on knees), the individual uses to sit and lift from the ground. Independent notes are assigned for each of the two acts - sit and stand up. The maximum grade is 5 for each of the two acts, one point being lost for each support or even half a point for any perceptible imbalance.
creatine kinase levels | six weeks
  U/l
Schober test | six weeks
  To check the mobility of the lumbar spine

CONTACTS AND LOCATIONS:
Overall Officials: Daniele MK Nardino, Specialist, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Rodrigo Antonio Carvalho ANDRAUS, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster C. Monitoring training in athletes with reference to overtraining syndrome. Med Sci Sports Exerc. 1998 Jul;30(7):1164-8. doi: 10.1097/00005768-199807000-00023. PMID 9662690
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Camargo VM, Martins Bdo C, Jardim C, Fernandes CJ, Hovnanian A, Souza R. Validation of a treadmill six-minute walk test protocol for the evaluation of patients with pulmonary arterial hypertension. J Bras Pneumol. 2009 May;35(5):423-30. doi: 10.1590/s1806-37132009000500006. English, Portuguese. PMID 19547850
- [Background] Abreu AM, Faria CD, Cardoso SM, Teixeira-Salmela LF. [The Brazilian version of the Fear Avoidance Beliefs Questionnaire]. Cad Saude Publica. 2008 Mar;24(3):615-23. doi: 10.1590/s0102-311x2008000300015. Portuguese. PMID 18327449
- [Background] Vigatto R, Alexandre NM, Correa Filho HR. Development of a Brazilian Portuguese version of the Oswestry Disability Index: cross-cultural adaptation, reliability, and validity. Spine (Phila Pa 1976). 2007 Feb 15;32(4):481-6. doi: 10.1097/01.brs.0000255075.11496.47. PMID 17304141
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Pimenta CA, Teixeiro MJ. [Proposal to adapt the McGill Pain Questionnaire into Portuguese]. Rev Esc Enferm USP. 1996 Dec;30(3):473-83. Portuguese. PMID 9016160
- [Derived] Nardin DMK, Stocco MR, Aguiar AF, Machado FA, de Oliveira RG, Andraus RAC. Effects of photobiomodulation and deep water running in patients with chronic non-specific low back pain: a randomized controlled trial. Lasers Med Sci. 2022 Jun;37(4):2135-2144. doi: 10.1007/s10103-021-03443-6. Epub 2022 Mar 4. PMID 35246766